CLINICAL TRIAL: NCT04074655
Title: Investigating the Effect of Training With a Virtual Reality Driving Simulator on Orientation Skills in Individuals With Some Memory Impairments
Brief Title: Investigating the Effect of Training With a Virtual Reality Driving Simulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019:073
Record Dates: First submitted 2019-08-26; First posted 2019-08-30 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2019-07

CONDITIONS: Spatial Navigation; Navigation, Spatial; Dementia
Keywords: Driving Simulator; Virtual Reality
MeSH Terms: conditions — Spatial Navigation; Dementia

STUDY DESIGN:
Intervention Model Description: In this study we do not need to label participants as healthy or demented; we only use the MoCA range between 7 to 25 to enroll participants. Many healthy adults do have some memory impairments and have a MoCA score less than 25 but still consider themselves healthy. Thus, we do not label anyone in this study as healthy or demented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Participants of the study will play the driving simulator daily (5 days/week) for 15-20 minutes/day over a period of 2 consecutive weeks.
  Interventions: Device: Driving Simulator in a Virtual Reality Environment

INTERVENTIONS:
Device: Driving Simulator in a Virtual Reality Environment — Driving simulator in virtual reality environment is a game with the several level of difficulty and the goal of improving the cognition level of participants in general and their spatial cognition in particular. Moreover this game, will have a positive effect on its users' mood as well.

SUMMARY:
The proposed study aims to investigate the use of a driving simulator in a virtual reality (VR) environment to improve the cognition state and spatial navigation of individuals with mild/moderate memory impairment.

All volunteers will be assessed by the Montreal Cognitive Assessment (MoCA),Montgomery-Asberg Depression Scale (MADRS) and Morris Water orientation tests for baseline assessment after they sign the consent form and are enrolled into the study. Participants will also be scheduled for post-intervention assessments (MADRS, Morris Water Orientation and a simple questionnaire on how they evaluate the experiment).

Participants of the study will play the driving simulator daily (5 days/week) for 15-20 minutes/day over a period of 2 consecutive weeks. Participants' daily performance data are recorded and uploaded on the secure server of the Priciple Investigator (PI).

Simulator Sickness Questionnaire (SSQ) test will also be run after the first session of the experiment and at the end of the training period.

DETAILED DESCRIPTION:
After obtaining their consent and enrolling into the study, participants of the study will commit themselves to use the driving simulator daily (5 days/week), and 15-20 minutes/day for a period of 2 consecutive weeks. The location for these simulation sessions will be one of the Family rooms of the Lindenwood Retirement Community. During the experiment, the research assistant (RA) of the study will be present and monitor participants for any plausible simulator sickness. In case if a participant presents any simulator sickness symptom, the experiment will be stopped and the RA will remain with the participant until s/he feels alright to go back to his/her room or with a caregiver. The RA and PI may withdraw the participant from the study if it is for their benefit.

Participants' performance data and the duration of which they practice are all being recorded and uploaded on the secure server of the PI. After the end of the 2-week exercise program, participants will be assessed again by Morris Water orientation test, SSQ, and MADRS; SSQ test will also be run after the first session of the experiment.

Furthermore, their feedback about using the driving simulator will be collected through a

ELIGIBILITY:
Inclusion criteria:

We will recruit up to 30 volunteers with mild/moderate memory impairment. Inclusion/Exclusion Criteria

* Age: 50+ years
* Have a score of 7< MoCA < 25
* Except the MCI/Alzheimer's diagnosis, have no known or diagnosis of major depression, bipolar disorder, schizophrenia, mood disorder, Parkinson's disease, Huntington disease, Amyotrophic Lateral Sclerosis (ALS), Multiple sclerosis (MS), and/or any other neurological disorder.
* Fluency in reading/understanding English

Furthermore, in this study we do not need to label participants as healthy or demented; we only use the MoCA range between 7 to 25 to enroll participants. Many healthy adults do have some memory impairments and have a MoCA score less than 25 but still consider themselves healthy. Thus, we do not label anyone in this study as healthy or demented.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
The ratio between the total trajectories and the trajectories in the correct quadrant (Morris water virtual reality test) | Baseline and Intervention (end of 2-week exercise)
  Spatial orientation virtual reality experiment equivalent to Morris water test as primary outcome measure.
  This test is one of the PI's team designs used in a previous study (B2016:073), which is the VR replica of the standard Morris Water test; and will be run at baseline and at the end of trial (post-intervention). In this test participants sit behind a computer monitor and they move within a virtual maze to reach a particular target. They will do this test using the laptop screen. The test has 5 trials, and participants' trajectory to reaching the target is recorded. The ratio between the total trajectories and the trajectories in the correct quadrant, quadrant of which the target is placed in, is reported as the error of participant trying to find the target.

SECONDARY OUTCOMES:
MADRS assessment | Baseline and Intervention (end of 2-week exercise)
  Montgomery-Asberg Depression Scale (MADRS) to measure depression as a confounding variable.
  The MADRS is a ten item rating scale for rating levels of depression. Each item is rated on a 7-point scale from 0 to 6, where 0 indicates absence of the symptom and 6 indicates extreme presence of the symptom. So, the maximum raw score of the test will be 60. The raw score reported more than 10, indicates the possible presence of depression. The time frame for the scale is the previous four weeks.
SSQ questionnaire | First session of the exercise and Intervention (end of 2-week exercise)
  Simulator Sickness Questionnaire (SSQ) to assess the plausible motion sickness due to using the driving simulator.
  The SSQ is a sixteen item questionnaire for rating the severity of most common symptoms associated with motion sickness, nausea and oculo-motor problems, experienced by users of virtual reality systems. Each item is rated on a 4-point scale from 0 to 3, where 0 indicates absence of the symptom and 3 indicates the symptom being severe. The total raw score reported by the questionnaire is 48, and the higher the reported score the more severe the symptoms experienced due to simulation sickness. The SSQ will be run after the first session of using the driving simulator and at the end of the trial (post-intervention).
Satisfaction questionnaire | Intervention (end of 2-week exercise)
  Short questionnaire to assess the level of satisfaction after using the driving simulator to collect participants' general feedback on the experiment.
  This is a short questionnaire consisting of 3 questions for rating the level of participants' satisfaction after using the driving simulator. Each item is rated on a 10-point scale from 1 to 10, representing from low to high satisfaction levels. The total raw score for the questionnaire is 30, and the higher the score, the higher the level of the satisfaction after using the driving simulator. This test will be run at the end of the trial (post-intervention).

CONTACTS AND LOCATIONS:
Locations (1):
- Lindenwood Manor, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Still has not been decided to share Individual Participant Data (IPD) with other researchers or not.

REFERENCES:
- [Derived] Masoumzadeh S, Moussavi Z. Does Practicing with a Virtual Reality Driving Simulator Improve Spatial Cognition in Older Adults? A Pilot Study. Neurosci Insights. 2020 Nov 3;15:2633105520967930. doi: 10.1177/2633105520967930. eCollection 2020. PMID 35174332